CLINICAL TRIAL: NCT06671249
Title: A Multicenter, Open and Prospective Randomized Controlled Trial Comparing the Safety and Cosmetic Outcomes of Laparoscopic Breast-conserving Surgery Versus Traditional Open Breast-conserving Surgery.
Brief Title: Comparing the Safety and Cosmetic Outcomes Between Laparoscopic Versus Traditional Open Breast-conserving Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1251
Record Dates: First submitted 2024-10-23; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic breast-conserving surgery (Experimental): Subjects who is going to accept laparoscopic breast-conserving surgery.
  Interventions: Procedure: Laparoscopic breast-conserving surgery
- Traditional open breast-conserving surgery (Active Comparator): Subjects who is going to accept traditional open breast-conserving surgery.
  Interventions: Procedure: Traditional open breast-conserving surgery

INTERVENTIONS:
Procedure: Laparoscopic breast-conserving surgery — Use laparoscopic surgery to treat breast cancer patients who want and have the opportunity to preserve their breast
  Arms: Laparoscopic breast-conserving surgery
Procedure: Traditional open breast-conserving surgery — Treat breast cancer patients who want and have the opportunity to preserve their breast with traditional open breast-conserving surgery.
  Arms: Traditional open breast-conserving surgery

SUMMARY:
In recent years, laparoscopic breast cancer surgery has received wide attention. It has advantages of minimal invasiveness, clear anatomical exposure, and good aesthetic effects. Based on these advantages, we propose whether laparoscopy is suitable for breast-conserving surgery for breast cancer. The standard procedure of laparoscopic breast-conserving surgery is unclear. More high-quality clinical studies are required. Therefore, we intend to conduct a multi-center, open, productive, randomized controlled study comparing the safety and cosmetic effects of endoscopic breast-conserving with traditional open breast-conserving surgery.

DETAILED DESCRIPTION:
In recent years, laparoscopic breast cancer surgery has received wide attention. It has advantages of minimal invasiveness, clear anatomical exposure, and good aesthetic effects. Based on these advantages, we propose whether laparoscopy is suitable for breast-conserving surgery for breast cancer. The standard procedure of laparoscopic breast-conserving surgery is unclear. More high-quality clinical studies are required to ensure the efficiency of cure. Also, less scars and breast preservation has becoming more and more important for patients' acceptance to the treatment. Therefore, we intend to conduct a multi-center, open, productive, randomized controlled study comparing the safety and cosmetic effects of endoscopic breast-conserving with traditional open breast-conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female over the age of 18
* Preoperative pathologically confirmed invasive breast cancer or ductal carcinoma in situ
* Clinical classification T1, T2 (maximum tumor diameter ≤5cm)
* Single-center tumor (preoperative confirmation by B-ultrasound, MRI and other imaging examinations)
* No clinical or imaging evidence of distant metastasis
* Able and willing to sign informed consent

Exclusion Criteria:

* Tumor in the lower inner quadrant
* Tumor in multiple quadrants
* Imaging or intraoperative pathology indicates tumor invasion of the nipple areola, skin, or pectoralis major
* Locally advanced breast cancer patients are undergoing neoadjuvant therapy
* Tumor in multiple quadrants
* Have been participating in other clinical trials, which may affect the participation in this trial
* Previous history of breast cancer (patients with recurrence after ipilateral breast-conserving surgery)
* Pregnant and lactating women
* Patients with severe cardiopulmonary disease or severely impaired lung function are not suitable for surgical establishment of an air cavity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
breast appearance satisfaction | 2 years
  Whether laparoscopic breast-conserving and traditional open breast-conserving had significant differences postoperative cosmetic outcomes. One of the evaluation indicators is breast appearance satisfaction. Our study chooses BREAST-Q questionnaire to evaluate patients' breast appearance satisfaction.
breast aesthetic scores | 2 years
  Whether laparoscopic breast-conserving and traditional open breast-conserving had significant differences postoperative cosmetic outcomes. Another of the evaluation indicators is breast aesthetic scores. We will invite two Plastic surgeons who did not participate in the study to judge patients' photographs, which is taken 18 months after the surgery, according to the Harris evaluation criteria.

SECONDARY OUTCOMES:
Complications | 1 year
  The study focus on intraoperative/postoperative complications between endoscopic breast-conserving and traditional open breast-conserving, including bleeding, hematoma, seroma, poor wound healing, nipple/areola necrosis, incision infection and incision dehiscence.
Quality of Life | 1 year
  Whether laparoscopic breast-conserving and traditional open breast-conserving have difference in quality of life. The study measures the quality of life with the EORTC QLQ BR23 questionnaire launched by European Organization for Research and Treatment of Cancer.
local recurrence rate | 2 years
  Whether laparoscopic breast-conserving and traditional open breast-conserving have difference in local recurrence rate. If local recurrence appears, record the time and location of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochen - Wang, Doctorate, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Xiaochen Wang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No